CLINICAL TRIAL: NCT05596643
Title: Investigation of Autonomic Dysfunction in Patients With Familial Mediterranean Fever
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2021.1427
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Familial Mediterranean Fever; Autonomic Dysfunction
Keywords: Familial Mediterranean Fever; Autonomic Dysfunction; r-r interval variability; sympathetic skin response
MeSH Terms: conditions — Familial Mediterranean Fever; Primary Dysautonomias | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients diagnosed with Familial Mediterranean Fever
  Interventions: Diagnostic Test: Composite Autonomic Symptom Score-31; Diagnostic Test: r-r interval variability with normal breathing; Diagnostic Test: r-r interval variability with deep breathing; Diagnostic Test: Valsalva ratio; Diagnostic Test: 30:15 ratio; Diagnostic Test: sympathetic skin response; Diagnostic Test: blood pressure response to standing; Diagnostic Test: blood pressure response to sustained handgrip test; Other: Hospital anxiety and depression scale; Diagnostic Test: Fibromyalgia rapid screening tool; Other: Familial Mediterranean Fever Quality of life scale; Other: Jenkins Sleep Evaluation Scale; Other: The Fatigue Severity Scale
- Healthy Controls
  Interventions: Diagnostic Test: Composite Autonomic Symptom Score-31; Diagnostic Test: r-r interval variability with normal breathing; Diagnostic Test: r-r interval variability with deep breathing; Diagnostic Test: Valsalva ratio; Diagnostic Test: 30:15 ratio; Diagnostic Test: sympathetic skin response; Diagnostic Test: blood pressure response to standing; Diagnostic Test: blood pressure response to sustained handgrip test; Other: Hospital anxiety and depression scale; Diagnostic Test: Fibromyalgia rapid screening tool; Other: Jenkins Sleep Evaluation Scale; Other: The Fatigue Severity Scale

INTERVENTIONS:
Diagnostic Test: Composite Autonomic Symptom Score-31 — Standardized questionnaire to determine the level of autonomic dysfunction
  Other Names: COMPASS-31
Diagnostic Test: r-r interval variability with normal breathing — electrophysiological test to detect parasympathetic dysfunction
Diagnostic Test: r-r interval variability with deep breathing — electrophysiological test to detect parasympathetic dysfunction
Diagnostic Test: Valsalva ratio — electrophysiological test to detect parasympathetic dysfunction
Diagnostic Test: 30:15 ratio — electrophysiological test to detect parasympathetic dysfunction
Diagnostic Test: sympathetic skin response — electrophysiological test to detect sympathetic dysfunction
  Other Names: SSR
Diagnostic Test: blood pressure response to standing — clinical test to detect sympathetic dysfunction
Diagnostic Test: blood pressure response to sustained handgrip test — clinical test to detect sympathetic dysfunction
Other: Hospital anxiety and depression scale — Standardized questionnaire to investigate the depression and anxiety
  Other Names: HADS
Diagnostic Test: Fibromyalgia rapid screening tool — Standardized questionnaire to determine the presence of fibromyalgia
  Other Names: FIRST
Other: Familial Mediterranean Fever Quality of life scale — Standardized questionnaire to investigate the quality of life in Familial Mediterranean Fever patients
  Other Names: FMFQoL
  Groups: Patients diagnosed with Familial Mediterranean Fever
Other: Jenkins Sleep Evaluation Scale — Standardized questionnaire to investigate the sleep quality and disturbance
Other: The Fatigue Severity Scale — Standardized questionnaire to investigate the fatigue severity
  Other Names: FSS

SUMMARY:
Familial Mediterranean Fever (FMF) is the most common inherited autoinflammatory disease affecting 150,000 patients worldwide. Periodic febrile exacerbations, peritonitis, and pleuritis are characteristic disease features. Dysregulation of IL-1β secretion has an important role in the pathophysiology of the disease, and IL-1β also serves as a therapeutic target. Chronic inflammation has been associated with early atherosclerotic and cardiovascular disease in various rheumatic diseases. An increased risk for cardiovascular events associated with disease activity has been described in rheumatoid arthritis, psoriatic arthritis, and systemic lupus erythematosus. In addition, autonomic nervous system dysfunction may contribute to increased cardiovascular risk in patients with inflammatory disease. For example, decreased heart rate variability is an important feature of cardiac autonomic dysfunction and is an isolated risk factor for cardiovascular events. Autonomic dysfunction studies related to FMF have conflicting results.

The aim of this study was to determine autonomic dysfunction symptoms and objective findings in patients with FMF; Demographic characteristics, disease characteristics, inflammatory burden, fatigue level, sleep quality, presence of fibromyalgia and their relationship with quality of life were evaluated and compared with healthy controls.

ELIGIBILITY:
Inclusion Criteria:

Familial Mediterranean Fever group;

1. Being between the ages of 18-65
2. Having a definite diagnosis of Familial Mediterranean Fever according to Livneh criteria

Healthy control group;

1. Being between the ages of 18-65
2. Absence of any disease diagnosis

Exclusion Criteria:

1. Liver or kidney failure
2. Pregnancy
3. Diabetes mellitus
4. Thyroid diseases
5. Those who use neuroprotective or antihypertensive drugs
6. Vitamin B12 deficiency
7. Anemia
8. Paraneoplastic neuropathy
9. Alcoholism
10. Cardiac failure
11. Cardiac arrhythmia
12. Acute thrombosis
13. Having a diagnosis of another systemic rheumatic disease
14. Persons who did not give consent to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with FMF Healthy control group
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Composite Autonomic Symptom Score-31 | 6 months
  It is a widely applicable, up-to-date, easy-to-apply and scientifically-based test that evaluates autonomic symptoms and functions by the person himself. It consists of 31 multiple-choice questions in 6 autonomic areas: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder function and pupillomotor areas. A score in the range of 0-100 is obtained as a result of multiplying each area by the weight factor determined by the study. High score indicates presence and severity of autonomic dysfunction.
r-r interval variability with normal breathing | 6 months
  The active and reference superficial recording electrodes are on the dorsal side of both hands, and the ground electrode is placed on the wrist. The R-R interval variability is calculated automatically by the electromyography device over a 1-minute recording.
r-r interval variability with deep breathing | 6 months
  The active and reference superficial recording electrodes are on the dorsal side of both hands, and the ground electrode is placed on the wrist. In order to determine the R-R interval variability with deep breathing, the patient is given 6 to 8 deep breaths, consisting of 5 seconds of inspiration followed by 5 seconds of expiration, and the result is automatically calculated by the electromyography device.
Valsalva ratio | 6 months
  The active and reference superficial recording electrodes are on the dorsal side of both hands, and the ground electrode is placed on the wrist. The test was performed by asking the subject to sit quietly and then blow into a mouthpiece attached to an aneroid pressure gauge at a pressure of 40 mmHg for 15 seconds. The ratio of the longest R-R interval shortly after the manoeuver (within about 20 beats) and the shortest R-R interval during the manoeuver is then measured. The result was expressed as the Valsalva ratio that is taken as the mean ratio from three successive Valsalva manoeuvers.
30:15 ratio | 6 months
  The active and reference superficial recording electrodes are on the dorsal side of both hands, and the ground electrode is placed on the wrist.The R-R interval on the ECG was recorded and used to determine the instantaneous HR at rest and then on the 15th and 30th beats after standing. The HR should normally rise after about 30 seconds as part of the response to return the blood pressure (BP) to normal. After standing up, the 30:15 ratio obtained by dividing the longest R-R distance around the 30th beat by the shortest R-R distance around the 15th beat was calculated automatically by the EMG device.
sympathetic skin response | 6 months
  Sweating that occurs in response to many different stimuli, electrolyte in the skin triggers changes in skin conductivity, resulting in instantaneous changes in skin conductivity. Sympathetic skin response evaluates these instantaneous changes in the skin in response to sweating. Sympathetic skin response reflects the function of sympathetic nerve fibers.Active recording electrodes on palm and sole; reference electrodes is placed on the back of the hand and the back of the foot. Responses obtained by applying electrical current over the median nerve trace are evaluated.
blood pressure response to standing | 6 months
  Participants were asked to stand up for 3 minutes after a 10-minute resting period in a supine position. The systolic and diastolic BP (SBP and DBP) just before standing, and 3 minutes after active standing were determined, in order to define postural change in BP and to evaluate orthostatic intolerance.
blood pressure response to sustained handgrip | 6 months
  Blood pressure measurement is continued at 1-minute intervals while patients perform sustained handgip at 30% of their maximum volitional strength for 5 minutes.The absolute difference between the highest DBP during handgrip and the basal DBP just before the handgrip was noted.

SECONDARY OUTCOMES:
Familial Mediterranean Fever Quality of Life Scale (FMF-QoL) | 6 months
  FMF-QoL was developed to evaluate the quality of life in FMF patients. This scale consists of 20 questions in the form of a Likert scale and the total scoring is between 0-80. High scores indicate a decrease in quality of life.
Hospital Anxiety and Depression Scale (HADS) | 6 months
  This scale consists of 14 questions in total, and anxiety symptoms are questioned in half of the questions and depression-related complaints in the other half. A subscore of 8 or higher for depression or anxiety is considered a clinical case.
Fibromyalgia Rapid Screening Tool (FIRST) | 6 months
  This scale consists of 6 questions investigating the most relevant clinical features of fibromyalgia. The questions are answered as yes/no and 5 or more out of 6 points in total are in favor of fibromyalgia.
The Fatigue Severity Scale (FSS) | 6 months
  It consists of a total of 9 questions in which complaints related to fatigue are scored between 0 and 7, taking into account the fatigue in the last week. The mean score is obtained by dividing the total score by 9, and it is defined as <4.0 points as no fatigue, 4.0-5.0 points at the border, and >5.0 points as fatigue.
Jenkins Sleep Evaluation Scale (JSS) | 6 months
  It is a scale in which scores between 0 and 5 are made for each symptom by questioning how many days in a month 4 sleep-related symptoms are experienced considering the last 1 month. The total score is between 0-20, and as the score increases, sleep quality deteriorates.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Tuncay Duruöz, Prof, Principal Investigator — Marmara University
Locations (1):
- Marmara University School of Medicine, Pendik Education and Research Hospital, Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No